CLINICAL TRIAL: NCT01916512
Title: Investigation of Relationship Between Cholesteryl Ester Transfer Protein Deficiency and Carotid/Coronary Atherosclerosis in Patients With Hyperalphalipoproteinemia
Brief Title: Relationship Between CETP Deficiency and Atherosclerosis in Patients With Hyperalphalipoproteinemia
Acronym: INFINITY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Osaka University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: INFINITY
Record Dates: First submitted 2013-07-22; First posted 2013-08-05 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2013-08

CONDITIONS: Low CETP Activity; CETP Deficiency; Hyperalphalipoproteinemia; Hyper-LDL-cholesterolemia; High Level of Remnant Cholesterol
Keywords: CETP, HDL, LDL, apoB-100, apoB-48, remnants
MeSH Terms: conditions — Cholesteryl Ester Transfer Protein Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine whether high high density lipoprotein-cholesterol(HDL-C) level and low Cholesteryl Ester Transfer Protein(CETP) activity is atherogenic or not in subjects who received health checkups. We investigate the association between CETP activities and the severity of atherosclerosis assessed by intima-media thickness (IMT) and compare the atherogenic change between in subjects with high HDL-C level, low HDL-C level, high CETP activities and low CETP activities by examining the morbidity rate of atherogenic diseases, the rate of ischemic electrocardiography(ECG) change, Calc Score of artery from chest X-ray, Ankle Brachial Index/Pulse Wave Velocity and various serum atherogenic markers. And we also examine the correlation between normal lipid profile and concentration, activity and function of surface lipoprotein in subjects with variety of lipoprotein levels, including patients with hyper-LDL-cholesterolemia, hyper-HDL-cholesterolemia with low or no CETP activity, patients with high level of remnant cholesterol or hyperlipoproteinemia of apolipoprotein(Apo)B-48.

ELIGIBILITY:
Inclusion criteria:

Subjects who are at the age of 40 and above and undergo annual health check in Omagari area including Daisen city and Yokote city and who provide written informed consent.

Exclusion criteria:

1. Those who do not provide written informed consent.
2. Those who are not able to take tests.
3. Those who are regarded not adequate as subject of this study by their physicians.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will explain about this study with the attached leaflet to the male and female examinees at the age of 40 and above who undergo annual health check up at Hiraga General Hospital in Akita Prefecture and obtain written consent to participate in the study. The written consents will be stored. The participant information will be made anonymous with sequential ID numbers. However the comparative lists of each participant and ID number will be stored in the locked shelf in case of disclosure requests from participants in future. The above will be conducted at Hiraga hospital and the samples will be sent to and measured to collect data in Osaka University. The analysis of data will be done at Osaka University and Akita University.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Difference of Ischemic changes of ECG among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of Ischemic changes of ECG was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of Calc Score of Aorta by Chest X-ray among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of Calc Score of Aorta by Chest X-ray was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of Ankle Brachial Index (ABI) among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of Ankle Brachial Index (ABI) was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of Pulse Wave Velocity (baPW) among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of Pulse Wave Velocity (baPW) was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of IMT and Plaque Score of Carotid artery among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of IMT and Plaque Score of Carotid artery was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of CETP activity between normolipidemic subjects and patients with dyslipidemia (including high HDL-C level) | participants will be followed for the duration of hospital stay（2 days）
  The difference of CETP activity was assessed between in those who do not satisfy any of these three conditions (normolipidemic subjects) and those who satisfy any of these three conditions (patients with dyslipidemia); LDL-C:100 mg/dl and above, HDL:80 mg/dl and above, TG:150 mg/dl and above.
Difference of Antioxidant activity between normolipidemic subjects and patients with dyslipidemia (including high HDL-C level) | participants will be followed for the duration of hospital stay（2 days）
  The difference of Antioxidant activity was assessed between normolipidemic subjects and patients with dyslipidemia;HDL from subjects' serum samples will be added to LDL with 2,2'-azobis(2-amidinopropane) dihydrochloride (AAPH).
Difference of Monocyte chemoattractant protein-1 (MCP-1) concentration between normolipidemic subjects and patients with dyslipidemia (including high HDL-C level) | participants will be followed for the duration of hospital stay（2 days）
  The difference of MCP-1 concentration was assessed between normolipidemic subjects and patients with dyslipidemia
Difference of Cholesterol efflux between normolipidemic subjects and patients with dyslipidemia (including high HDL-C level) | participants will be followed for the duration of hospital stay（2 days）
  The difference of Cholesterol efflux by HDL from macrophage was assessed between normolipidemic subjects and patients with dyslipidemia
Difference of Proteome analysis of lipoproteins between normolipidemic subjects and patients with dyslipidemia (including high HDL-C level) | participants will be followed for the duration of hospital stay（2 days）
  The difference of Proteome analysis of lipoproteins (HDL, LDL, remnant binding protein) was assessed between normolipidemic subjects and patients with dyslipidemia

SECONDARY OUTCOMES:
Difference of Fasting blood glucose and HbA1c among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of Fasting blood glucose and HbA1c was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of waist circumference among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of waist circumference was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of Smoking habits, alcohol taking habits and fitness habits among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of Smoking habits, alcohol taking habits and fitness habits was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of BMI among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of BMI was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of Blood Pressure among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of Blood Pressure was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of 75g glucose tolerance test and calculated homeostasis model assessment of insulin resistance (HOMA-IR) among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of 75g glucose tolerance test and calculated homeostasis model assessment of insulin resistance (HOMA-IR) was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of Total Cholesterol(TC) among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of Total Cholesterol(TC) was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of low density lipoprotein-cholesterol (LDL-C) among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of low density lipoprotein-cholesterol (LDL-C) was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of triglyceride (TG) among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of triglyceride (TG) was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of Serum adiponectin among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference ofSerum adiponectin was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of Apolipoprotein (apo)B-48 concentrations among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of Apolipoprotein (apo)B-48 concentrations was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of Remnant lipoprotein (RemL-C) among subjects with low/high CETP mass/activity and HDL-C level | participants will be followed for the duration of hospital stay（2 days）
  The difference of Remnant lipoprotein (RemL-C) was assessed between in subjects with high CETP mass/activity and in those with low CETP mass/activity, and between in subjects with high HDL-C level and in those with low HDL-C level
Difference of Lipoprotein Profile between normolipidemic subjects and patients with dyslipidemia (including high HDL-C level) | participants will be followed for the duration of hospital stay（2 days）
  The difference of Lipoprotein Profile analyzed by high performance liquid chromatography(HPLC) method was assessed between in those who do not satisfy any of these three conditions (normolipidemic subjects) and those who satisfy any of these three conditions (patients with dyslipidemia); LDL-C:100 mg/dl and above, HDL:80 mg/dl and above, TG:150 mg/dl and above.
Difference of apolipoprotein(apo)B-48 concentrations between normolipidemic subjects and patients with dyslipidemia (including high HDL-C level) | participants will be followed for the duration of hospital stay（2 days）
  The difference of apoB-48 concentrations was assessed between in normolipidemic subjects and in patients with dyslipidemia
Difference of Remnant lipoprotein (RemL-C) between normolipidemic subjects and patients with dyslipidemia (including high HDL-C level) | participants will be followed for the duration of hospital stay（2 days）
  The difference of RemL-C was assessed between in normolipidemic subjects and in patients with dyslipidemia

CONTACTS AND LOCATIONS:
Overall Officials: Shizuya Yamashita, MD, PhD, FAHA, FJCC, Study Chair — Osaka University Graduate School of Medicine; Etsuko Fushimi, MD, PhD, Study Director — Hiraga General Hospital; Hiroshi Itoh, MD, PhD, Study Director — Akita University Graduate School of Medicine; Norimichi Nakajima, MD, Study Director — Nakajima Naika Clinic; Yoshinobu Ikeda, MD, Study Director — Ikeda Clinic; Yuji Matsuzawa, MD, PhD, Study Director — Sumitomo Hospital
Locations (1):
- Osaka University Graduate School of Medicine, Suita, Osaka, Japan